CLINICAL TRIAL: NCT04789655
Title: A Phase 1, Multi-center, Open-label, Dose Finding Study of CC-96191 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of CC-96191 in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-96191-AML-001; U1111-1264-5412 (Registry Identifier: WHO); 2022-500573-13-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-09 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid
Keywords: Acute Myeloid Leukemia; CC-96191; Relapsed or refractory
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-96191 (Experimental): CC-96191 will be administered intravenously on a 28-day Cycle
  Interventions: Drug: CC-96191

INTERVENTIONS:
Drug: CC-96191 — CC-96191

SUMMARY:
This Phase 1, clinical study of CC-96191 will explore the safety, tolerability and preliminary biological and clinical activity of CC-96191 as a single-agent in the setting of Relapsed or refractory acute myeloid leukemia (R/R AML).

The dose escalation (Part A) of the study will explore escalating intravenous doses of CC-96191 to estimate the MTD and/or RP2D of CC-96191 as monotherapy.

The expansion (Part B), will further evaluate the safety and efficacy of CC-96191 administered at or below the MTD in one or more expansion cohorts in order to determine the RP2D.

ELIGIBILITY:
Inclusion Criteria

* Participants must satisfy the following criteria to be enrolled in the study:.
* Participant must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
* Participant is ≥ 18 years of age at the time of signing the ICF.
* Relapsed or refractory CD33 positive AML at last visit as defined by the World Health Organization (WHO) Classification who have failed or who are ineligible for or have refused all available therapies for AML which may provide clinical benefit.
* Participant has Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* At least 4 weeks (from first dose) has elapsed from donor lymphocyte infusion without conditioning.
* Females and males must practice true abstinence or agree to contraceptive methods throughout the study, and during the safety follow-up period.

Exclusion Criteria

* The presence of any of the following will exclude a Participant from enrollment:.
* Participant is suspected or proven to have acute promyelocytic leukemia (FAB M3) based on morphology, immunophenotype, molecular assay, or karyotype.
* Participant has received systemic anticancer therapy (including investigational therapy) or radiotherapy < 28 days or 5 half-lives, whichever is shorter, prior to the start of study treatment. Hydroxyurea is allowed to control peripheral leukemia blasts.
* Participants with prior autologous hematopoietic stem cell transplant who, in the investigator's judgment, have not fully recovered from the effects of the last transplant (eg, transplant-related side effects).
* Prior allogeneic HSCT with either standard or reduced intensity conditioning ≤ 6 months prior to dosing.
* Participants on systemic immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). The use of topical steroids for ongoing skin or ocular GVHD is permitted.
* Participant has persistent, clinically significant non-hematologic toxicities from prior therapies which have not recovered to < Grade 2.
* Participant has or is suspected of having central nervous system (CNS) leukemia. Evaluation of cerebrospinal fluid is only required if CNS involvement by leukemia is suspected during screening.
* History of concurrent second cancers requiring active, ongoing systemic treatment.
* Participant is known seropositive or active infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus or hepatitis C virus.
* Impaired cardiac function or clinically significant cardiac diseases, as defined in the protocol.
* Participant is a pregnant or lactating female.
* Participant with isolated extramedullary disease without bone marrow involvement.
* Inadequate pulmonary function as defined as oxygen saturation (SpO2) < 92% on room air.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to 42 days after the first dose
  Are defined as toxicities that meet the protocol-specified criteria occurring within the DLT assessment window (Cycle 1, Days 1 to at least 28 and up to 42 days) that cannot be attributed to a clearly identifiable cause such as underlying illness, disease progression, other concurrent illness, or concomitant medication.
Maximum tolerated dose (MTD) | Up to 35 days after the last dose
  Is defined as the highest dose at which less than 33% of the population treated with CC-96191 experience a dose limiting toxicity (DLT) in the first cycle.
Adverse Events (AEs) | Up to 35 days after the last dose
  Type, frequency, seriousness, severity and relationship of AEs to CC-96191

SECONDARY OUTCOMES:
Complete remission rate (CRR) | Up to approximately 2 years
  As defined by the European Leukemia Net (ELN) AML response criteria.
Objective response rate (ORR) | Up to approximately 2 years
  As defined by the European Leukemia Net (ELN) AML response criteria.
Progression-free survival (PFS) | Up to approximately 2 years
  Is defined as the time from the first dose of CC-96191 to the first occurrence of disease progression or death from any cause.
Overall survival (OS) | Up to approximately 2 years
  Is measured as the time from the first dose of CC-96191 to death due to any cause.
Duration of remission | Up to approximately 2 years
  For subjects with best response of complete remission (CR) of any type, morphologic leukemia free state (MLFS) or partial remission (PR), duration of response (DOR) is measured from the time when criteria for CR/MLFS/PR are first met (whichever is first recorded) until the first date at which relapse, or progressive disease is objectively documented
Time to remission | Up to approximately 2 years
  Time from the date of first dose to the earliest date of any response (CR of any type, MLFS or PR)
Pharmacokinetics - Cmax | Up to 35 days after last dose
  Maximum serum concentration of drug
Pharmacokinetics - AUC | Up to 35 days after last dose
  Area under the serum concentration time-curve
Pharmacokinetics - tmax | Up to 35 days after last dose
  Time to peak (maximum) serum concentration
Pharmacokinetics - t1/2 | Up to 35 days after last dose
  Terminal half-life
Pharmacokinetics - CL | Up to 35 days after last dose
  Total body clearance of the drug from the serum
Pharmacokinetics - Vss | Up to 35 days after last dose
  Volume of distribution at steady-state
Presence of anti-drug antibodies (ADA) | Up to 35 days after last dose
  Detection of anti-drug antibodies in participants
Frequency of anti-drug antibodies (ADA) | Up to 35 days after last dose
  Frequency of anti-drug antibodies in participants

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (8):
  - Local Institution - 109, Birmingham, Alabama
  - Local Institution - 105, Jacksonville, Florida
  - Local Institution - 108, Atlanta, Georgia
  - Local Institution - 110, Rochester, Minnesota
  - Local Institution - 101, Hackensack, New Jersey
  - Local Institution - 102, New York, New York
  - Local Institution - 107, Houston, Texas
  - Local Institution - 111, Seattle, Washington
- Canada (2):
  - Local Institution - 202, Calgary, Alberta
  - Local Institution - 201, Toronto, Ontario
- France (4):
  - Local Institution - 303, Marseille
  - Local Institution - 304, Paris
  - Local Institution - 301, Pessac
  - Local Institution - 302, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Lunn-Halbert MC, Laszlo GS, Erraiss S, Orr MT, Jessup HK, Thomas HJ, Chan H, Jahromi MA, Lloyd J, Cheung AF, Chang GP, Dichwalkar T, Fallon D, Grinberg A, Rodriguez-Arboli E, Lim SYT, Kehret AR, Huo J, Cole FM, Scharffenberger SC, Walter RB. Preclinical Characterization of the Anti-Leukemia Activity of the CD33/CD16a/NKG2D Immune-Modulating TriNKET(R) CC-96191. Cancers (Basel). 2024 Feb 22;16(5):877. doi: 10.3390/cancers16050877. PMID 38473239
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com